CLINICAL TRIAL: NCT06214442
Title: Effects of Menstrual Cycle Phases on Plantar Flexor Neuromechanical Properties and Achilles Tendon Mechanical Properties of Eumenorrheic Women and Hormonal Contraception Users
Brief Title: Effects of the Menstrual Cycle on Triceps Surae Properties in Women
Status: Recruiting | Type: Observational
Sponsor: Marco Aurélio Vaz, PhD (Other)
Responsible Party: Sponsor-Investigator, Marco Aurélio Vaz, PhD, Principal Investigator, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Other Study IDs: 5.989.983
Record Dates: First submitted 2023-10-24; First posted 2024-01-19 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Menstrual Cycle; Achilles Tendon
Keywords: mechanical properties; material properties; morphological properites; estrogen; progesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Physically active eumenorrheic women with regular menstrual cycle: Women who practice physical exercise and have regular menstruation ranging from 25 to 38 days.
  Interventions: Other: Evaluations of the mechanical properties of the achilles tendon in different phases of the menstrual cycle
- Sedentary eumenorrheic women with regular menstrual cycle: Women who do not practice physical exercise and have regular menstruation ranging from 25 to 38 days.
  Interventions: Other: Evaluations of the mechanical properties of the achilles tendon in different phases of the menstrual cycle
- Physically active women using hormonal contraceptives: Physically active women using oral hormonal contraception combined with estrogen and progesterone within the last six months.
  Interventions: Other: Evaluations of the mechanical properties of the achilles tendon in different phases of the menstrual cycle
- Sedentary women who use hormonal contraception: Sedentary women using oral hormonal contraception combined with estrogen and progesterone within the last six months.
  Interventions: Other: Evaluations of the mechanical properties of the achilles tendon in different phases of the menstrual cycle

INTERVENTIONS:
Other: Evaluations of the mechanical properties of the achilles tendon in different phases of the menstrual cycle — Monitoring assessments to verify the effect of different phases of the menstrual cycle on the neuromechanical properties of the Achilles tendon.

SUMMARY:
The menstrual cycle is an important biological rhythm, whereby large cyclic fluctuations in endogenous sex hormones, such as estrogen and progesterone, are observed, which can affect performance. Evidence shows that endogenous and exogenous changes in hormone concentrations during the menstrual cycle exert many effects on the nervous and endocrine systems, in addition to the connective tissue, with consequences for the movement system. Pre-clinical studies (i.e., in animal models) show an estrogen association with the structural and mechanical properties of tendons and ligaments. Several elegant studies performed with female participants have tried to establish the mechanism underlying the effect of estrogen on collagen synthesis and its effects on exercise and functionality. Their findings suggest that the tendon properties may be affected when exposed to varying concentrations of estrogen. The largest tendon in humans, the Achilles tendon, has a direct role in functional capacity, activities of daily living, and locomotion. Studies show that the triceps surae's structural and mechanical properties may change throughout the menstrual cycle, and that these changes are related to endogenous and exogenous fluctuations in estrogen and progesterone. Musculotendinous stiffness, which is dependent on the collagen content, has been seen to vary considerably over the course of the menstrual cycle. In addition, it has been reported that females who have been taking the contraceptive pill for at least a year demonstrate lower levels of tendon strain compared to non-pill taking females, indicating a possible influence of hormonal state on tendon mechanical properties. However, the different experimental designs, the varied approaches to the evaluations and the lack of studies with high methodological quality limit our understanding of the effects of the different phases of the menstrual cycle on the triceps surae's neuromechanical properties. The aim of this observational study will be to investigate whether the morphological, mechanical (active and passive), material, and functional properties of the plantar flexor muscles and of the Achilles tendon, as well as functional parameters, change during voluntary contractions throughout the phases of the menstrual cycle in eumenorrheic women and in users of hormonal contraception. Understanding the acute effects of these properties in eumenorrheic women and users of hormonal contraception is essential so that we can adequately plan interventions and prescriptions of physical exercise and rehabilitation aimed for women.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the group of eumenorrheic women

  * Being eumenorrheic with a regular menstrual cycle lasting between 21 and 35 days during the last 6 months prior to study participation.
  * Body Mass Index between 20 and 25 kg/m2.
  * Normal ankle function and range of motion.
  * Do not use hormonal contraception of any kind or supplements hormones for at least the 6 months prior to the study.
  * No complaints of pain or history of lower limb injury.
  * In view of the COVID-19 pandemic, have completed vaccination will be used as an inclusion criteria.
  * For the physically active group, practice regular physical exercise at least 3 times a week for the past 6 months.
  * For the sedentary group, not practicing regular physical exercise in the last 6 months.

Inclusion criteria for the group users of hormonal oral contraception:

* Body Mass Index between 20 and 25 kg/m2.
* Normal ankle function and range of motion.
* Make use of any method of oral hormonal contraception (compressed).
* Make use of combined oral hormonal contraception with estrogen and progesterone (ethinylestradiol + Drospirenone) for at least 6 months before participating in the study.
* Do not use other hormone supplements for at least 6 months prior to the study.
* No complaints of pain or presence of pathologies in the lower limb
* In view of the COVID-19 pandemic, have completed vaccination will be used as an inclusion criteria.
* For the physically active group, practice regular physical exercise at least 3 times a week for the past 6 months.
* For the sedentary group, not practicing regular physical exercise in the last 6 months

Exclusion Criteria:

Exclusion Criteria for eumenorrheic and contraception hormonal groups:

Health problems - contraindication to maximal effort exercise. Additionally, the following subjects will be excluded:

* Women who have anovulatory cycles or phase lutea deficiency.
* Women in early menopause.
* Pregnant or lactating women.
* Women with oligomenorrhea (menstrual cycles longer than 35 days, or delay of menstruation for the same period).
* Women with hypothalamic amenorrhea.
* Female smokers.
* Women with metabolic syndrome.
* For women using hormonal contraceptives, women who use adhesive, injectable, intrauterine devices, implants, vaginal rings, as well as progesterone-only CH methods.
* Does not meet the inclusion criteria.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Over the last three decades, there has been a rise in the number of women participating in exercise, from physical activity to elite sports. However, the number of studies regarding female participants' performance is still small compared to male participants. The menstrual cycle is an important biological rhythm, whereby large cyclic fluctuations in endogenous sex hormones, such as estrogen and progesterone, are observed, which can affect performance.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal voluntary isometric contraction (Nm) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Maximal voluntary isometric contraction (MVIC) of the plantar flexor muscles, i.e., largest plantar flexor torque generated in different phases of menstrual cycle and different moments of contraception use
Achilles tendon stiffness (N/mm) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Achilles tendon stiffness will be calculated during maximal voluntary contraction in different phases of menstrual cycle and contraception users

SECONDARY OUTCOMES:
Cross-sectional area (mm²) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  The evaluation of the cross-sectional area will be carried out using ultrasound, evaluating proximal, medial and distal portions from the calcaneus bone.
tendon stress (MPa) during maximal voluntary contractions | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  The stress will be obtained by taking the ratio between Achilles tendon strength and tendon cross sectional area, and tension taking the relationship between tendon elongation and tendon length at rest
Myotendinous junction displacement (mm) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  The displacement of the myotendinous junction of the medial gastrocnemius muscle (DTJM) will be evaluated during passive torque assessment.The analysis will be carried out in three core cycles of the five passive torque cycles.
Ankle functionality (cm) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Ankle functionality and ankle dorsiflexion range of motion assessed through functional heel raise theses.
Blood concentrations (pg/ml) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Blood concentrations of estrogen and progesterone in different phases of menstrual cycle
Transvaginal ultrasound (cm) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Transvaginal ultrasound will be evaluated to control the menstrual cycle and take measurements of the ovary and uterus in the different phases of the menstrual cycle.
Tendon length (mm²) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  The length of the tendon will be assessed using ultrasound, starting from the myotendinous junction to the calcaneus bone. The measurement will be carried out with a measuring tape.
Strain (%) during maximal voluntary contractions | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  strain will be evaluated through the relationship relationship between tendon deformation and tendon length at rest. ratio between tendon elongation and TL at rest.
Hysteresis (%) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Hysteresis measurements will be obtained from five cycles, but they will begin at 30° of plantar flexion, and the ankle will be passively moved until maximum dorsal flexion that is achieved. Both passive torque and hysteresis will be evaluated at a constant angular velocity of 5°.s
Passive torque (Nm) | The assessment will be performed at the beginning (1-4 days), middle (10-14 days), and end (22-26 days) of Cycle 1 (each menstrual cycle is between 28-30 days).
  Passive torque will be evaluated with the isokinetic method dynamometer moving the ankle passively for five cycles, from 0° (i.e. 90° angle between foot and leg) to the maximum ROM previously determined for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vaz, Study Chair — Federal University of Rio Grande do Sul; Marco Vaz, Study Director — Federal University of Rio Grande do Sul; Marco Vaz, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Marco Aurelio Vaz, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: No